CLINICAL TRIAL: NCT04657445
Title: EFFECT OF COVID-19 DISEASE IN SMELL AND TASTE OF PATIENTS WITH MILD, MODERATE OR SEVERE SYMPTOMATOLOGY
Status: Completed | Type: Observational
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Liontos Angelos, CONSULTANT OF INTERNAL MEDICINE, University Hospital, Ioannina
Other Study IDs: 931/17-11-2020
Record Dates: First submitted 2020-12-06; First posted 2020-12-08 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Olfactory and Taste Dysfunction in SARS-CoV2 Infection
Keywords: Olfactory, taste dysfunction, SARS-CoV2, COVID-19
MeSH Terms: conditions — Anosmia; Taste Disorders; COVID-19 | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- home-quarantined patients: home-quarantined patients
  Interventions: Diagnostic Test: visual analogue scale
- inhospitalized patients: inhospitalized patients
  Interventions: Diagnostic Test: visual analogue scale

INTERVENTIONS:
Diagnostic Test: visual analogue scale — A visual analog scale (VAS) is a measurement device used to quantify a subjective experience.

SUMMARY:
This is an observational data and recording study. The aim of our study is to investigate the effect of SARS-COV2 infection on patients' sense of smell and taste, through quality control measurements using optic analogue scale (VAS) in hospitalized and in home-quarantined patients.

DETAILED DESCRIPTION:
Eligible participants who will be recruited in this research protocol will be adult patients who are diagnosed positive for SARS-COV2, infection with Real Time Polymerase Chain Reaction Test (RT-PCR).

The study population will be divided in two groups. The first group will be consisted with positive patients that were referred to either the Emergency Department (ED) of Infectious Diseases or at the Outpatient Clinic screening for SARS-COV2 and are being self-quarantined at home. The participants will be hospitalized patients in the Infectious Diseases Unit (IDU) of the University General Hospital of Ioannina.

The examination will be performed at the moment of diagnosis both for self-quarantine patients and for in hospitalized patients. The follow up evaluation will be a re-examination, performed at least four weeks after the moment of diagnosis. The time internal of reassessing the patients chosen according to current literature, estimated that is the minimum reassessment interval and seems to be a reference time for either progression stabilization or recession of the symptoms of anosmia/ ageusia (12, 13).

Patients will be asked to evaluate their olfactory and gustatory abilities through the visual analogue scale (VAS), at three time points: 1.before infection( as they can recall it), 2. at the time of diagnosis and 3. four weeks later(14).

Patients' scoring will be recorded in a horizontal presentation of 100 VAS points, where zero refers to no smell or taste while 100 refers to normal sensation. In addition, patients will rate their nasal obstruction and rhinorrhea on a similar VAS scale, where 0 refers to a completely blocked nose and an excessively runny nose while 100 indicates normal nasal breathing and a no runny nose. All patients will assess the intensity of the olfactory and taste function, through a self testing them at home. Patients will rate from 0 to 100 the intensity of smell, after being exposed to five common household odors (ie lemon juice, oregano, instant coffee, toothpaste and mint gum).The choice of these substances is based on their influence at the irritation of the trigeminal nerve.

The intensity of taste function will be evaluated using four(4) substances: sugar, salt, lemon juice and instant coffee (decaffeinated), that represent the following 4 basic quality flavors:sweet, salty, sour and bitter. Every patient will have to receive orally half a teaspoon of each testant and report the quality of taste perception. After each testant they have to rinse their mouth with tap water. Bitter testant will have to be tested in the end.

Patient demographics, associated symptoms, and comorbidities will be recorded. The patients will have to report and fill in symptoms such as fever, cough, shortness of breath or dyspnea, fatigue, muscle aches, runny nose, blocked nose, loss of smell, and loss of taste.

The results will be recorded in a questionnaire.

Covid-19 positive patients recovering at home, will be informed for the study either by telephone or in person, following all the safety measures provided by National Organization of Public Health of Greece, by one of the investigators officially participating in the study. A questionnaire will be completed by the examinee, after telephone information about the purpose of the study and after providing a written consent from.

In hospitalized patients in the Infectious Diseases Unit, will be informed by the investigators participating in the study and will follow the above procedure.

This study was submitted for approval to the research ethic committee and the scientific council of University General Hospital of Ioannina and was accepted.

ELIGIBILITY:
Inclusion Criteria:

* adult>18 years old

  * COVID-19 positive patient, via RT-PCR test
  * Patient referred to the University General Hospital of Ioannina

Exclusion Criteria:

* Age <18

  * Previous nasal surgery, endoscopic sinus surgery
  * Head and neck radiotherapy
  * Head injury
  * Allergic rhinitis
  * Chronis Rhinosinusitis
  * Psychiatric/ Neurological disorders
  * Disorders that altering the level of consciousness (Glasgow Coma Scale <15)
  * History of smell and taste disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be divided in two groups. The first group will be consisted with positive patients that were referred to either the Emergency Department (ED) of Infectious Diseases or at the Outpatient Clinic screening for SARS-COV2 and are being self-quarantined at home. The participants of the second group will be hospitalized patients in the Infectious Diseases Unit (IDU) of the University General Hospital of Ioannina.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
oflactory and taste dysfunction in SARS-CoV2 infection | 4 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: CHARALAMPOS MILIONIS, PROFESSOR, Principal Investigator — University Hospital, Ioannina; IOANNIS KASTANIOUDAKIS, PROFESSOR, Principal Investigator — University Hospital, Ioannina
Locations (1):
- University General Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: No